CLINICAL TRIAL: NCT03564899
Title: The Breast Cancer & Physical Activity Level (BC-PAL) Pilot Study
Acronym: BC-PAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Christine Friedenreich, Principal Investigator, AHS Cancer Control Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BC-PAL
Record Dates: First submitted 2018-05-29; First posted 2018-06-21 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer Survivorship
Keywords: Breast cancer; Survivorship; Physical activity intervention; Activity trackers; Sedentary time
MeSH Terms: conditions — Breast Neoplasms; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomized, using a 1:1:1 allocation, into one of three groups: 1) the control group (no physical activity intervention), 2) the lighter intensity physical activity intervention or 3) the higher intensity physical activity intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): Receive no physical activity intervention (maintain baseline physical activity participation)
- Lighter intensity physical activity (Experimental): Receive an intervention of 300 minutes/week of physical activity at an intensity of 40-60% of heart rate reserve for 12 weeks.
  Interventions: Behavioral: Lighter intensity physical activity intervention
- Higher intensity physical activity (Active Comparator): Receive an intervention of 150 minutes/week of physical activity at an intensity of 60-80% of heart rate reserve for 12 weeks.
  Interventions: Behavioral: Higher intensity physical activity intervention

INTERVENTIONS:
Behavioral: Lighter intensity physical activity intervention — Prescription of 300 minutes/week of physical activity at an intensity of 40-60% of heart rate reserve
  Arms: Lighter intensity physical activity
Behavioral: Higher intensity physical activity intervention — Prescription of 150 minutes/week of physical activity at an intensity of 60-80% of heart rate reserve
  Arms: Higher intensity physical activity

SUMMARY:
The Breast Cancer & Physical Activity Level (BC-PAL) pilot study is a randomized controlled pilot trial aimed at evaluating whether total physical activity levels, health-related fitness and patient reported outcomes are improved by promoting different intensities of physical activity participation within a home-based setting, and whether these improvements are maintained over the long-term, in inactive breast cancer survivors.

DETAILED DESCRIPTION:
Detailed Description

Rationale and Significance:

Breast cancer is the most common cancer among Canadian women. Physical activity has emerged as a potential lifestyle factor for improving rehabilitation and survival after breast cancer. The American Cancer Society recommends that cancer survivors engage in at least 150 minutes of moderate-vigorous intensity physical activity per week. However, only ≈ 15% of breast cancer survivors reported meeting these physical activity guidelines. Therefore, interventions that promote physical activity behavior change in an unsupervised/home-based setting are needed to provide the necessary tools and support for breast cancer survivors. No study to date has assessed the effects of a lighter intensity physical activity intervention, compared to no additional physical activity prescription (control) or a higher intensity physical activity intervention (comparable to current exercise guidelines), in inactive breast cancer survivors, in addition to the longer-term maintenance effects of these interventions.

Study Aims:

Aim 1: To evaluate the effects of prescribing an additional 300 minutes/week of lighter intensity physical activity (LIPA) or 150 minutes/week of higher intensity physical activity (HIPA) versus no physical activity intervention (control) on total physical activity and sedentary time in inactive breast cancer survivors.

Aim 2: To evaluate the effects of prescribing an additional 300 minutes/week of LIPA or 150 minutes/week of HIPA versus control on markers of health-related fitness (anthropometric measures, body composition, cardio-respiratory fitness) and patient reported outcomes (quality of life, sleep quality, feelings of happiness, perceived feelings of depression) in inactive breast cancer survivors.

Aim 3: To evaluate the longer-term (24-week) maintenance effect of prescribing an additional 300 minutes/week of LIPA or 150 minutes/week of HIPA versus control on our primary and secondary outcomes.

Research Plan:

A three-armed, 12-week pilot randomized controlled trial followed by a 12-week follow-up measurement is proposed. All eligible and interested women are invited to contact and meet with study staff at the Holy Cross Center in Calgary, at which time the study protocol is explained, informed consent obtained and baseline questionnaires distributed. These questionnaires assess: demographic characteristics, sleep quality, perceived health-related quality of life, feelings of happiness and perceived feelings of depression. At the end of this first meeting, participants are asked to wear an Actigraph GTX3® accelerometer for seven days to assess baseline physical activity levels. During a second meeting at the Holy Cross Center, accelerometers are returned to study staff, anthropometric data (height, weight, waist and hip circumferences and body composition) are collected and a maximal treadmill test (modified Balke protocol) is conducted. Participants are then randomized, using a 1:1:1 allocation, into either the control (no intervention), lighter intensity or the higher intensity physical activity interventions. The control group is instructed to maintain baseline physical activity participation. The lighter intensity physical activity (LIPA) group is instructed to accumulate 300 minutes/week of physical activity at an intensity of 40-60% of heart rate reserve. The higher intensity physical activity (HIPA) group is instructed to accumulate 150 minutes of physical activity at an intensity of 60-80% of heart rate reserve. Participants randomized to the LIPA and HIPA groups are given: 1) instructions on physical activity safety and goal setting, proper heart rate monitoring and stretching techniques that should be completed before and after physical activity participation; 2) a publicly-available physical activity guidebook for breast cancer survivors; 3) a Polar A360® device to track heart rate and physical activity time throughout the intervention. Data collected by this device are uploaded to the Polar Flow® application by syncing with a smart phone or a computer with a provided USB cord. Participants are asked to upload their data at least once per week. If a participant does not own a computer or a smart phone, or prefers that the study staff upload these data for them, in-person meetings are arranged to do so. Participants in the LIPA and HIPA groups are also asked to rate the feasibility of achieving the prescribed physical activity targets and record strategies used and barriers encountered during the intervention in a diary. In-person/telephone meetings with these participants occur every three weeks to review data from the Polar A360® device and diary, to reinforce progress/good adherence and discuss/solve any problems or barriers to achieving the prescribed physical activity goals. During weeks 12 (final intervention week) and 24 (final week of the follow-up period), all participants wear an Actigraph GTX3® accelerometer to assess physical activity volume. At the end of weeks 12 (end of the intervention) and 24 (end of the follow-up period), all participants repeat baseline measurements and questionnaires, except for items on demographic characteristics.

The investigators will use intention-to-treat statistical analysis on all participants with follow-up data regardless of adherence to the interventions. An analysis of covariance (ANCOVA) will be used to compare between-group differences in study outcomes at 12- and 24-weeks, compared to baseline, after adjusting for baseline outcomes values.

This pilot randomized controlled trial will provide data on the feasibility of prescribing different physical activity intensities within a home-based setting to increase total physical activity time, reduce sedentary time and improve health outcomes in breast cancer survivors. The investigators will use these data to help design and conceptualize a larger-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed Stage I-III breast cancer diagnosis
* Completion of adjuvant treatment (chemotherapy, radiation therapy and surgery) except for hormone therapy
* Females ≥18 years of age
* Currently living in the Calgary area and able to meet with study staff at the Holy Cross Center on at least six occasions (twice as baseline, 12- and 24-weeks)
* Currently inactive (accumulating ≤ 60 minutes of moderate-vigorous intensity physical activity/week and ≤ 10,000 steps/day)
* Ability to undertake a physical activity program [assessed by an Exercise Physiologist with the Physical Activity Readiness Questionnaire (PAR-Q+)].

Exclusion Criteria:

* Deemed too active (accumulating on average ≥ 60 minutes of moderate-vigorous intensity physical activity/week and ≥ 10,000 steps/day)
* Being away from Calgary or not able to attend testing sessions/be contacted by study staff for > 4 consecutive weeks during the intervention period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in sedentary time, light intensity physical activity time and moderate-vigorous intensity physical activity time (hours/day) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Measured with accelerometry over seven days

SECONDARY OUTCOMES:
Change in body weight (kg) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Measured with a standard beam scale
Change in height (cm) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Measured with a stadiometer
Change in waist and hip circumference (cm) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Measured with an anthropometric measuring tape
Change in body composition (fat and lean mass in kg) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Measured by Dual X-ray Absorptiometry (DXA)
Change in cardiorespiratory fitness (VO2max) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Measured by maximal cardiorespiratory fitness test using the multistage, modified Balke treadmill protocol
Change in body mass index (BMI in kg/m2) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Weight and height will be combined to report BMI

OTHER OUTCOMES:
Change in sleep quality (scale of 0 to 21) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  Pittsburgh Sleep Quality Index will be used to measure the total aggregate score from the questionnaire on a scale of 0-21, with 21 indicating worst sleep quality
Change in health-related quality of life (scale of 0 to 100) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  The Medical Outcomes Study Short Form-12 Survey will be used to measure mental component aggregate score and physical component aggregate score, each on a scale of 0-100, with a higher score indicating higher function, well-being or quality of life. The questions on physical functioning, role-physical limitations and bodily pain are summed to provide the physical aggregate score. The questions on social functioning, vitality, role-emotional limitations and mental health are summed to provide the mental aggregate score.
Change in breast cancer-specific quality of life (scale of 0 to 28) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  The Functional Assessment of Cancer Therapy-Breast Questionnaire will be used to measure total score ranges from 0 to 28, with a higher score indicating higher function, well-being or quality of life. The results from each question are summed to provide the total score.
Changes in feelings of happiness (scale of 1 to 11 and value in % over past 7 days) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  The Happiness Scale will be used to assess happiness with one question asking participants what is the average level of happiness over the past 7 days on a scale of 1 (extremely happy) to 11 (extremely unhappy). A second question asks participants what is the percentage of time spent happy (value in % over the last 7 days), neutral (value in % over the last 7 days) and unhappy (value in % over the last 7 days).
Changes in perceived feelings of depression (scale from 0 to 27) | Baseline, 12 weeks (end of intervention) and 24 weeks (end of follow-up period)
  The Patient Health Questionnaire provides a score of 0 to 27, with a higher score indicating higher feelings of depression. The results from each question are summed to provide the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Friedenreich, PhD, Principal Investigator — CancerControl Alberta; Jessica McNeil, PhD, Study Director — CancerControl Alberta
Locations (1):
- The Rehabilitation, Exercise and Complementary (REACH) center within the Holy Cross Center, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McNeil J, Fahim M, Stone CR, O'Reilly R, Courneya KS, Friedenreich CM. Adherence to a lower versus higher intensity physical activity intervention in the Breast Cancer & Physical Activity Level (BC-PAL) Trial. J Cancer Surviv. 2022 Apr;16(2):353-365. doi: 10.1007/s11764-021-01030-w. Epub 2021 Mar 22. PMID 33754246
- [Derived] McNeil J, Brenner DR, Stone CR, O'Reilly R, Ruan Y, Vallance JK, Courneya KS, Thorpe KE, Klein DJ, Friedenreich CM. Activity Tracker to Prescribe Various Exercise Intensities in Breast Cancer Survivors. Med Sci Sports Exerc. 2019 May;51(5):930-940. doi: 10.1249/MSS.0000000000001890. PMID 30694978